CLINICAL TRIAL: NCT05097963
Title: A Prospective Study of Endoscopic Ultrasound Shear Wave Elastography for Assessment of Liver Fibrosis
Brief Title: A Study to Evaluate Liver Stiffness With Shear Wave Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinay Chandrasekhara, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-003779
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Liver Disease; Advanced Fibrosis; Advanced Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects undergoing EUS shear wave elastography (Experimental): Subject who are eligible will undergo EUS for clinical indications. EUS shear wave measurements will be gathered and studied to determine diagnostic accuracy when compared to MR Elastography.
  Interventions: Device: Endoscopic Ultrasound Shear Wave Elastography

INTERVENTIONS:
Device: Endoscopic Ultrasound Shear Wave Elastography — Software to determine stiffness of liver for evaluating liver fibrosis.

SUMMARY:
The purpose of the study is to assess the diagnostic accuracy of Endoscopic Ultrasound (EUS) shear wave elastography in liver fibrosis staging in both normal subjects and subjects with advanced liver fibrosis/cirrhosis

DETAILED DESCRIPTION:
This is a prospective, paired study. Study subjects who are scheduled to undergo EUS at Mayo Clinic will be identified through Epic. Chart review will be performed including review of prior imaging, medical history, and laboratory results as available in Epic to determine study eligibility. Subjects without history of chronic liver disease (screened by low FIB-4 score) and those with known advanced fibrosis/cirrhosis will be eligible for the study. Eligible study subjects will then be contacted either before, or at the time of their endoscopy procedure to discuss study participation. All subjects will then receive standard clinical care based on the indication for the EUS procedure. During the EUS procedure, study subjects with undergo shear wave measurements obtained in a non-invasive manner as part of the endosonographic evaluation of the liver. 10 measurements (including shear wave velocity (Vs), elastic modulus (E)) will be obtained for point SWE (pSWE). Measurements will be obtained from both left and right lobes of liver unless technically infeasible to do so. Study subjects will then undergo a paired MR elastography (same day or at later date) after completion of EUS and only if consistent and reliable shear wave measurements were obtained (e.g., VsN > 70%(reliability index of each measurement expressed in percentages), IQR/M (interquartile range/ Median) is <15% for Vs and <30% for E). Enrolled study subjects who had undergone a previous MRE (within 6 months of enrollment) would be eligible for the study, without the need to undergo further research MRE. After completion of MR elastography, the subjects will then continue through their routine clinical care and will not be followed up by research staff. The expected duration of subject participation is anticipated to begin at the time of study enrollment and terminate after completion of MR elastography. There will be no additional follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age who are undergoing EUS procedures.
* Subjects with history of chronic liver disease, advanced fibrosis or cirrhosis
* Subjects without any history of chronic liver disease
* Subjects who underwent MR elastography within six (6) months of enrollment will be eligible to participate in the study.
* Subjects able to give appropriate consent to the study or have an appropriate representative to do so.

Exclusion Criteria:

* Subjects who may have MRI-incompatible metal implants/devices.
* Subjects with severe claustrophobia who may not tolerate MR elastography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Termite F, Borrelli de Andreis F, Liguori A, Gasbarrini A, Attili F, Spada C, Miele L. The Role of Endoscopic Ultrasound in Assessing Portal Hypertension: A State-of-the-Art Literature Review and Evolving Perspectives. Liver Int. 2025 Apr;45(4):e16176. doi: 10.1111/liv.16176. Epub 2024 Nov 27. PMID 39601324
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- EUS Shear Wave Elastography: Subjects who underwent EUS for clinical indications. EUS shear wave measurements were gathered and studied to determine diagnostic accuracy when compared to Magnetic Resonance (MR) Elastography.
  Endoscopic Ultrasound Shear Wave Elastography: Software to determine stiffness of liver for evaluating liver fibrosis.
Period: Overall Study
Arm/Group | EUS Shear Wave Elastography
Started | 63
Completed | 29
Not Completed | 34
Not completed — Protocol Violation | 13
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Groups:
- EUS Shear Wave Elastography: Subjects who underwent EUS for clinical indications. EUS shear wave measurements were gathered and studied to determine diagnostic accuracy when compared to MR Elastography.
  Endoscopic Ultrasound Shear Wave Elastography: Software to determine stiffness of liver for evaluating liver fibrosis.
Arm/Group | EUS Shear Wave Elastography
Number analyzed (Participants) | 63
Age, Continuous [Mean (Full Range); unit: years] | 52 [30 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Median Endoscopic Ultrasound (EUS) Shear Wave Elastography
Description: EUS shear wave elastography accuracy obtained by Elastic modulus measurements automatically calculated and a median of 10 readings is generated. Measured as kilopascals (kPA)
Time Frame: baseline
Population: Data was not collected or analyzed for 34 subjects.
Measure: Median (Full Range); unit: kPA
Arm/Group | EUS Shear Wave Elastography
Number analyzed (Participants) | 29
kPA | 0.11 [0.05 to 0.17]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 1 day
Arm/Group | EUS Shear Wave Elastography
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT05097963/Prot_SAP_000.pdf